CLINICAL TRIAL: NCT05756465
Title: The Effect of Smartphone-Based Virtual Reality Relaxation (S-VR) On the Comfort on Cancer Patients Undergoing Chemotherapy: A Randomized Controlled Trial
Brief Title: The Effect of Smartphone-Based Virtual Reality Relaxation (S-VR) in Cancer Patients Undergoing Chemotherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gadjah Mada University (Other)
Collaborators: Taipei Medical University (Other)
Responsible Party: Principal Investigator, Made Satya Nugraha Gautama, Principal Investigator, Master of Nursing Program, Faculty of Medicine, Public Health, and Nursing Universitas Gadjah Mada, Gadjah Mada University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 12117
Record Dates: First submitted 2023-01-22; First posted 2023-03-06 (Actual); Last update posted 2024-06-24 (Actual); Status verified 2024-06

CONDITIONS: Comfort; Pain; Anxiety; Blood Pressure; Pulse Rate
Keywords: Immersive virtual reality; Comfort; Cancer patient; Chemotherapy
MeSH Terms: conditions — Pain; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: This study is a two-arm parallel randomised controlled trial with a 1:1 allocation. This study divided two groups, namely the intervention group in the form of SVR therapy with the installation of a VR device (head-mounted display/HMD) on the respondent's head during chemotherapy. The control group received standard care through leaflets containing instructions for relaxation techniques with image visualization as guided imagery therapy. The group's determination, apart from randomization, will also use envelope concealment and outcome assessor will be blinded during data collection. The protocol is composed according to Standard Protocol Items: Recommendations for Interventional Trials and its checklist
Who Masked: Outcomes Assessor
Masking Description: Outcome assessor (Nurse who appointed by researcher to be responsible for collection of outcome data) and data analysts will be blinded from participant allocation. This blinding is carried out, due to the technical nature of VR interventions, making it difficult to blind study participant during the intervention, thus to minimize the potential for methodological bias, the study must blind the outcome assessor or data analysts.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SVR group (Experimental): Participant in the intervention arm will receive immersive virtual reality intervention in the form of VR box (Shinecon 6.0 VR Box Virtual Reality Glasses with headphones). SVR is virtual relaxation and distraction therapy through a smartphone-based VR device (head-mounted display) which attached to the head of cancer patient during chemotherapy, by displaying a virtual environment of natural panoramas in 360-degree video and combined with traditional and classic musical audio instruments (non-copyright).
  Interventions: Device: Smartphone-based virtual reality relaxation (SVR)
- Control group (No Intervention): In the control group, participants will be given standard care in the form of guided imagery leaflets. It is an information sheets in the form of leaflets about the meaning, benefits, and ways of doing guided imagery relaxation therapy for cancer patient during chemotherapy. RA will guide the participants to practice the guided imagery relaxation therapy listed on the leaflet for ± 10 minutes.

INTERVENTIONS:
Device: Smartphone-based virtual reality relaxation (SVR) — SVR is virtual relaxation and distraction therapy through a smartphone-based VR device (head-mounted display) that is attached to the head of a cancer patient undergoing chemotherapy, displaying a virtual environment of natural panoramas in 360-degree video and combined with traditional and classic musical instruments. SVR device is paired with smartphone using operating system either Android (minimum generation 11, Android 4.4 KitKat) or OS version 12, minimum screen size of 5.5-inch and maximum of 6.0-inch, screen resolution of at least 1080 x 1920 pixels, can connect to WIFI/ internet and provides a YouTube app to access 360-degree videos. SVR content uses original 360o videos produced by researchers using a video editor software for ± 10 minutes duration.
  Arms: SVR group

SUMMARY:
The aim of this trial study is to identify the effect of S-VR on comfort on cancer patients undergoing chemotherapy. Additional objectives of this study include: (a) identifying the effect of S-VR on anxiety in chemotherapy patients; (b) identifying the effect of S-VR on pain intensity of chemotherapy patients; (c) identifying the effect of S-VR on vital signs (pulse and blood pressure) of chemotherapy patients. Participants is randomly assigned into two group: SVR intervention group and control group. In the SVR group, participants will use a VR device (head-mounted display/HMD) with 360-degree natural panoramic and music relaxation contents. Control group will receive standard care in the form of guided imagery leaflet.

The research will adhere to the ethical standards outlined in the Declaration of Helsinki and its subsequent amendments, as well as the protocol under reviewed by Medical and Health Research Ethics Committee (MHREC) Faculty of Medicine, Public Health and Nursing Universitas Gadjah Mada - Dr. Sardjito General Hospital Yogyakarta (Approval Number: KE/FK/0301/EC/2023). A formal informed consent will be obtained from all study participants. Validation number: 63f81182672f3 (http://komisietik.fk.ugm.ac.id/validasi)

DETAILED DESCRIPTION:
This study presents Smartphone-Based Virtual Reality Relaxation (S-VR) as a complementary modality in cancer treatment. We will conduct a randomised controlled trial to evaluate its impact in cancer patient undergoing chemotherapy.

This study is a two-arm parallel randomised controlled trial with a 1:1 allocation. This study divided two groups, namely the intervention group in the form of SVR therapy with the installation of a VR device (head-mounted display/HMD) on the respondent's head during chemotherapy. The control group received standard care through leaflets containing instructions for relaxation techniques with image visualization as guided imagery therapy. The group's determination, apart from randomization, will also use envelope concealment and outcome assessor will be blinded during data collection. The protocol is composed according to Standard Protocol Items: Recommendations for Interventional Trials and its checklist.

The sample size calculation used the G*Power for windows application Version 3.1.9.6. The effect size is 0.81, type 1 error (α) = 5% (two-tailed), power (1-β) 90%, and the allocation ratio between groups is 1:1. Effect size refers to previous studies with similar outcomes. Based on the G Power calculation, the calculation of study sample size is 34 people per group. We will drop out by 15%, thereby increasing the sample size to 40 subjects per group.

The sampling technique will use consecutive sampling. This non-probability sampling method involves recruiting everyone from the accessible population during a given time interval or for a specific sample size. Cancer patients who have scheduled chemotherapy and meet the requirements in the data collection time will be offered to be involved in the study.

Researchers will carry out the screening process to determine eligible patients as study participants. The patient's medical record will also be validated to fulfill the baseline information (e.g. anthropometric data, laboratory, patient identification, and laboratory result). Allocation sequence generation will be through simple randomization of study participant using a formulation from the Microsoft Excel program (randbetween formula) and allocation sequence concealment will use sealed envelope. Participants in the intervention and control groups will be treated with concealment from received envelopes containing random numbers from the randomization procedure. Outcome assessor (Nurse who appointed by researcher to be responsible for collection of outcome data) and data analysts will be blinded from participant allocation. This blinding is carried out, due to the technical nature of VR interventions, making it difficult to blind study participant during the intervention, thus to minimize the potential for methodological bias, the study must blind the outcome assessor or data analysts.

Patients who are scheduled for chemotherapy will go through an assessment stage (such as checking the latest laboratory results, medical records, vital signs, and electrocardiogram results) by the nurse on duty to determine if they are eligible and pass the screening to go to the chemotherapy session. Then, patients who pass the screening will be asked about their willingness to be involved and fill the informed consent. Patients who are willing (signed informed consent) will be given a sealed envelope. The envelope will contain random numbers for group allocation. Firstly, participants will be evaluated (pre-test) by the outcome assessor (research nurse) in the same room before entering the chemotherapy room. After the evaluation is complete, the researcher will open the envelope of the participants and see the random numbers obtained (without the participants' knowledge and the outcome assessor). If the numbers obtained are in the order of numbers 1 - 40, then participants will be directed to the chemotherapy room on the east side (intervention group); otherwise, if they get numbers 41 - 80, they will be directed to the chemotherapy room on the west side (control group). A research assistant (RA) will accompany each room. We will arrange and place the intervention and control groups in different chemotherapy rooms, with each research assistant will accompany the group to minimize contamination of information both between participants, participants and intervention providers, between intervention providers, intervention providers, and nurses or doctors on duty.

Participant in the intervention arm will receive immersive virtual reality intervention in the form of VR box (Shinecon 6.0 VR Box Virtual Reality Glasses with headphones). SVR is virtual relaxation and distraction therapy through a smartphone-based VR device (head-mounted display) which attached to the head of cancer patient during chemotherapy, by displaying a virtual environment of natural panoramas in 360-degree video and combined with traditional and classic musical audio instruments (non-copyright). SVR device is paired with smartphone using operating system either Android (minimum generation 11, Android 4.4 KitKat) or OS version 12, minimum screen size of 5.5-inch and maximum of 6.0-inch, screen resolution of at least 1080 x 1920 pixels, can connect to WIFI/ internet and provides a YouTube app to access 360 degree videos. SVR content uses original 360-degree videos produced by researchers using a video editor software for ± 10 minutes duration. The duration was determined based on previous study, where this duration may be effective in anticipating patient saturation related to content and preventing motion sickness. 360-degree video is created directly with chosen at panoramic views of Yogyakarta, Indonesia and Taipei, Taiwan. RA will provide information and introduce SVR intervention for approximately 5 minutes, help pair the SVR devices to the patient and start the intervention for approximately 10 minutes.

In the control group, participants will be given standard care in the form of guided imagery leaflets. It is an information sheets in the form of leaflets about the meaning, benefits, and ways of doing guided imagery relaxation therapy for cancer patient during chemotherapy. RA will guide the participants to practice the guided imagery relaxation therapy listed on the leaflet for ± 10 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Cancer patients are receiving chemotherapy in all cycles.
* Age ≥ 18 years.
* Performance status (ECOG Score) 0 - 2.
* Ability to understand and sign the informed consent

Exclusion Criteria:

* Cancer patients with a history of skull structures or cervical spine abnormalities that complicate using VR devices.
* Cancer patients with cognitive, visual and hearing impairment, wearing glasses, or having chemo - port.
* Patients with a history of epilepsy, seizures, drug and/or drug addiction, vertigo, or visually induced motion sickness.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2023-03-27 (Actual); Primary Completion 2023-05-30 (Actual); Study Completion 2023-07-30 (Actual)

PRIMARY OUTCOMES:
the Shortened General Comfort Questionnaire | Change from baseline the Shortened General Comfort Questionnaire at immediately after one session of chemotherapy (regardless of drug administration duration)
  Subjective responses of cancer patients during one session of chemotherapy administration (regardless of how many chemotherapy cycles, for instance in the first cycle, second cycle and so on) in four dimensions of comfort including physical, social, psychospiritual, and environmental are measured using a questionnaire. It measure using the Shortened General Comfort Questionnaire in Indonesian version. The questionnaire consists of 28 statement items with a Likert scale and an assessment score from 1 (strongly disagree) to 6 (strongly agree). The highest total score from the comfort instrument is 168 and the lowest is 28. The higher scores indicate higher level of comfort.

SECONDARY OUTCOMES:
Evaluation of Anxiety | T0: Baseline data collection T1: 10 minutes before chemotherapy premedication; T2: 10 minutes before start the intervention; T3: immediately after received intervention; T4: 60 minutes after drugs administration is completed.
  Transitory emotional reactions of cancer patients that arise in situations during one session of chemotherapy administration (regardless of how many chemotherapy cycles, for instance in the first cycle, second cycle and so on) which is perceived as threatening, were measured using a questionnaire. It is measured using the Visual Analog Scale for Anxiety (VAS - A). The scale consisted of a 100-mm horizontal line, embedded on the left by the words ''not at all anxious'' and on the right by ''extremely anxious.'' A higher score indicated greater anxiety.
Evaluation of Pain | T0: Baseline data collection T1: 10 minutes before chemotherapy premedication; T2: 10 minutes before start the intervention; T3: immediately after received intervention; T4: 60 minutes after drugs administration is completed.
  Cancer patients' unpleasant sensory and emotional sensations occur during one session of chemotherapy administration (regardless of how many chemotherapy cycles, for instance in the first cycle, second cycle and so on) due to cancer diagnosis, invasive procedures, and acute side effects of cytotoxic agents. It is measured using the Numerical Rating Pain Scale (NPS). Pain intensity items are scored using an 11-point numeric rating scale. A higher score indicated greater pain.
Evaluation of Pulse rate | T0: Baseline data collection T1: 10 minutes before chemotherapy premedication; T2: 10 minutes before start the intervention; T3: immediately after received intervention; T4: 60 minutes after drugs administration is completed.
  Pulse rate is a measurement of the heart rate, or the number of times the heart beats per minute in cancer patients before intravenous access, before receiving the intervention, immediately after the intervention, and after one session of chemotherapy administration is completed. Adults' regular resting heart rate ranges from 60 to 100 beats per minute. It is measured by using automatic digital sphygmomanometer.
Evaluation of Blood pressure (systolic blood pressure and diastolic blood pressure) | T0: Baseline data collection T1: 10 minutes before chemotherapy premedication; T2: 10 minutes before start the intervention; T3: immediately after received intervention; T4: 60 minutes after drugs administration is completed.
  Blood pressure is as objective measurement are measured by using automatic digital sphygmomanometer. BP is the force exerted by circulating blood against the walls of the body's arteries, the main blood vessels in the body in cancer patients who will be given intravenous access, before receiving the intervention, immediately after the intervention, and after one session of chemotherapy administration is completed. A systolic pressure above 90 mm Hg and less than 120 mm Hg, and a diastolic pressure between 60 mm Hg and less than 80 mm Hg.

CONTACTS AND LOCATIONS:
Overall Officials: Made Satya Nugraha N Gautama, Master, Principal Investigator — Gadjah Mada University
Locations (2):
- Indonesia (2):
  - Universitas Gadjah Mada, Sleman, Special Region of Yogyakarta
  - Dr Sardjito General Hospital, Yogyakarta

IPD SHARING:
Plan to Share IPD: No
All information relating to the identity of the research subject will be kept confidential by the researcher. The results of this study will be published without mentioning the identity of the research subject.

REFERENCES:
- [Background] Fabi A, Fotia L, Giuseppini F, Gaeta A, Falcicchio C, Giuliani G, Savarese A, Taraborelli E, Rossi V, Malaguti P, Giannarelli D, Pugliese P, Cognetti F. The immersive experience of virtual reality during chemotherapy in patients with early breast and ovarian cancers: The patient's dream study. Front Oncol. 2022 Sep 30;12:960387. doi: 10.3389/fonc.2022.960387. eCollection 2022. PMID 36249001
- [Background] Bilgic S, Acaroglu R. Effects of Listening to Music on the Comfort of Chemotherapy Patients. West J Nurs Res. 2017 Jun;39(6):745-762. doi: 10.1177/0193945916660527. Epub 2016 Aug 11. PMID 27515501
- [Background] Chan AW, Tetzlaff JM, Gotzsche PC, Altman DG, Mann H, Berlin JA, Dickersin K, Hrobjartsson A, Schulz KF, Parulekar WR, Krleza-Jeric K, Laupacis A, Moher D. SPIRIT 2013 explanation and elaboration: guidance for protocols of clinical trials. BMJ. 2013 Jan 8;346:e7586. doi: 10.1136/bmj.e7586. PMID 23303884
- [Background] Faul F, Erdfelder E, Buchner A, Lang AG. Statistical power analyses using G*Power 3.1: tests for correlation and regression analyses. Behav Res Methods. 2009 Nov;41(4):1149-60. doi: 10.3758/BRM.41.4.1149. PMID 19897823
- [Derived] Gautama MSN, Haryani H, Huang TW, Chen JH, Chuang YH. Effectiveness of smartphone-based virtual reality relaxation (SVR) for enhancing comfort in cancer patients undergoing chemotherapy: a randomized controlled trial. Support Care Cancer. 2024 Nov 26;32(12):824. doi: 10.1007/s00520-024-09036-7. PMID 39589559
- [Derived] Gautama MSN, Haryani H, Huang TW. Efficacy of smartphone-based virtual reality relaxation in providing comfort to patients with cancer undergoing chemotherapy in oncology outpatient setting in Indonesia: protocol for a randomised controlled trial. BMJ Open. 2023 Jul 25;13(7):e074506. doi: 10.1136/bmjopen-2023-074506. PMID 37491084